CLINICAL TRIAL: NCT03013140
Title: Pre-optimization of Fluid Status to Prevent Hypotension by Non-invasive Arterial Pressure Monitor During Cesarean Section
Brief Title: Preloading to Prevent Hypotension During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201610025RIND
Record Dates: First submitted 2016-12-22; First posted 2017-01-06 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2019-07

CONDITIONS: Obstetric Anesthesia Problems
Keywords: Anesthesia, Obstetric; fluid therapy; cesarean section; spinal anesthesia
MeSH Terms: interventions — Fluid Therapy; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Goal-directed preloading (Experimental): Fluid therapy: Within 30 minutes before spinal anaesthesia, repeat "Ringer's Injection" 3ml/kg within 3 minutes with 1-min gap until change in SV (ΔSV) <5%
  Interventions: Drug: Fluid therapy; Procedure: Spinal anaesthesia
- Preloading (Active Comparator): Fluid therapy: Within 30 mins before spinal anaesthesia, infuse 1000ml "Ringer's injection" with a pressurizer within 15 minutes.
  Interventions: Procedure: Spinal anaesthesia

INTERVENTIONS:
Drug: Fluid therapy — Goal directed Fluid therapy: Within 30 minutes before spinal anaesthesia, repeat "Ringer's Injection" 3ml/kg within 3 minutes with 1-min gap until ΔSV<5%
  Other Names: "Ringer's Injection"
  Arms: Goal-directed preloading
Procedure: Spinal anaesthesia — Inject marcaine and fentanyl to CSF for anaesthesia

SUMMARY:
Whether the usage of non-invasive arterial blood pressure monitor to guide fluid therapy in caesarean section can effectively reduce the incidence of hypotension and fetal complications.

DETAILED DESCRIPTION:
Spinal anesthesia in the cesarean section often causes significant peripheral vascular dilatation, decreases blood pressure and cardiac output reduction which leads to maternal nausea, vomiting, dizziness and uteroplacental hypoperfusion. Infusion therapy and the use of vasopressor can prevent and treat the incidence of hypotension. Appropriate fluid therapy can not only maintain maternal tissue perfusion, but also reduce uteroplacental hypoperfusion. In the present study, perioperative goal directed fluid therapy is used. The non-invasive continuous hemodynamic monitor is used in this study, and the parameters (blood pressure (BP), stroke volume(SV), stroke volume variation (SVV), cardiac output (CO)) are used to determine the parameters of the blood transfusion in cesarean section as infusion guidelines. The application of Clearsight system to the pre-infusion of target-guided crystalloid solution is compared with the infusion of quantitative crystalline solution in the hope of reducing the incidence of maternal hypotension, reducing the use of vasopressin, improving uteroplacental perfusion and reducing the incidence of fetal acidosis.

ELIGIBILITY:
Inclusion criteria:

1. 20-45 y/o parturient
2. Receive spinal anesthesia (SA) or combined spinal-epidural anesthesia (CSA) to undergo cesarean section

Exclusion criteria:

1. Emergent C/S
2. BMI>35kg/m2
3. Height <150cm or >175 cm
4. Patients with major cardiovascular disease, preeclampsia or eclampsia.
5. Gestational age < 36wks
6. Multiple pregnancy

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2019-06-09 (Actual)

PRIMARY OUTCOMES:
Incidence of maternal hypotension | delivery

SECONDARY OUTCOMES:
Dosage of vasopressor | delivery
Total fluid volume | delivery

CONTACTS AND LOCATIONS:
Overall Officials: YiShiuan Lin, Principal Investigator — National Taiwan University Hospital
Locations (1):
- NTUH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang SH, Lin YS, Lee CN, Cheng YJ, Chen YH, Chiu HC, Wu CY. Implications of Continuous Noninvasive Finger Cuff Arterial Pressure Device Use during Cesarean Delivery for Goal-Directed Fluid Therapy Preload Optimization: A Randomized Controlled Trial. Biomed Res Int. 2021 Mar 28;2021:6685584. doi: 10.1155/2021/6685584. eCollection 2021. PMID 33855080